CLINICAL TRIAL: NCT00674713
Title: Effect of Acupuncture on Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Germano De Cosmo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1014/05
Record Dates: First submitted 2008-05-05; First posted 2008-05-08 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Cholelithiasis
Keywords: Patients undergoing laparoscopic cholecystectomy for cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Acupuncture Therapy; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- A (Experimental): Patients receiving acupuncture at P6 point plus physiological saline solution
  Interventions: Other: Acupuncture; Drug: Physiological saline solution
- B (Active Comparator): Patients receiving ondansetron plus sham acupuncture
  Interventions: Drug: Ondansetron; Other: Sham acupuncture
- C (Other): Patients receiving ondansetron plus acupuncture at P6 point
  Interventions: Drug: Ondansetron; Other: Acupuncture at P6 point
- D (Placebo Comparator): Patients receiving physiological saline solution plus sham acupuncture
  Interventions: Drug: Physiological saline solution; Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture
  Arms: A
Drug: Ondansetron
  Arms: B
Drug: Physiological saline solution
  Arms: A
Other: Sham acupuncture
  Arms: B
Drug: Ondansetron
  Arms: C
Other: Acupuncture at P6 point
  Arms: C
Drug: Physiological saline solution
  Arms: D
Other: Sham acupuncture
  Arms: D

SUMMARY:
The aim of the study is to investigate if P6 acupuncture made after induction of general anaesthesia might be effective for the prevention of PONV as ondansetron and if the acupuncture-ondansetron combination could enhance single therapy efficacy in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I-II scheduled for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patient's refusal
* Patients with history of carpal tunnel syndrome or eczema at P6 point
* Pregnant patients
* Female patients in a phase of the menstrual cycle other than premenstrual, nausea and vomiting within 24 hours before anaesthesia
* Known allergy to anti-inflammatory drugs, opioids and ondansetron.
* Patients with a pre-existing chronic pain disorder or with a gastrointestinal disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Germano De Cosmo, MD, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy